CLINICAL TRIAL: NCT02442895
Title: Predictors of Ovarian Response in Women Undergoing Ovarian Stimulation for IVF
Brief Title: Biomarkers of Ovarian Reserve and Correlation With IVF Treatments
Status: Completed | Type: Observational
Sponsor: U.O.S. Procreazione Medicalmente Assistita e Congelamento Gameti (Other)
Responsible Party: Principal Investigator, Dr.ssa Raffaella Depalo, Director of U.O.S. Procreazione Medicalmente Assistita e Congelamento Gameti, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, U.O.S. Procreazione Medicalmente Assistita e Congelamento Gameti
Other Study IDs: Uospmacg2
Record Dates: First submitted 2015-04-27; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Pregnancy, Ovarian
Keywords: mature oocytes; antral follicles count; follicle stimulating hormone; antimullerian hormone
MeSH Terms: conditions — Pregnancy, Ovarian

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Long luteal protocol: Subcutaneous administration of GnRH agonist (Triptorelina pamoato 0.1 mg/ml) in the medium-luteal phase (21th day) of the cycle before the stimulation. The next menstruation, in the presence of estradiol level (E2)<30pg/ml and in the absence of follicular cysts, the gonadotropin stimulation was begun. In the presence of at least three follicles of diameter ≥18mm was induced final oocyte maturation by administration of human chorionic gonadotropin (hCG).
- Daily antagonist protocol: GnRH antagonist (cetrorelix acetate 0.25 mg) was administered subcutaneously with a fixed protocol from the day +6 of stimulation or with a flexible protocol from the day in which at least one follicle reached a diameter of 14mm. In both protocols GnRH antagonist was administered until the day of the assumption of hCG. Recombinant Follicle Stimulating Hormone (rFSH) was administered from the 3rd day of menstruation at a dose of 150-300 IU/die according to the characteristics of women. The hCG was administered when at least three follicles had reached 18 mm in diameter and estradiol levels were higher than 150 pg/mL/dominant follicle.
- Depot antagonist protocol: GnRH antagonist (Cetrorelix acetate 0.25 mg) was administered subcutaneously with a fixed or flexible protocol until the day of the assumption of hCG. Corifollitropila alfa was used at dose of 100μg (in women with weight ≤60 kg and age ≤36 years) or 150μg (in women with weight> 60 kg of any age or weight ≥50 kg and age greater than 36 years). Corifollitropina alfa was administered subcutaneously in the day +3 and in the day +5 or +6 was supplemented with rFSH at doses 112-300 IU/day.
  The hCG was administered when at least three follicles had reached 18 mm in diameter and estradiol levels were higher than 150 pg/mL/dominant follicle.

SUMMARY:
Retrospective study to evaluate the correlation between AFC, FSHb, AMH and IVF outcomes of 347 cycles performed with three different protocols.

DETAILED DESCRIPTION:
347 IVF cycles (236 patients) analyzed for a retrospective study to evaluate the correlation between the biomarkers of ovarian reserve (antral follicles count, antimullerian hormone, basal follicle stimulating hormone) and number of oocytes and mature oocytes (MII) retrieved during the pick up. For the stimulation were used three different protocols: long luteal, antagonist with daily administration of gonadotropins and antagonist with depot administration of gonadotropins.

ELIGIBILITY:
Inclusion Criteria:

* women with primary or secondary infertility underwent ovarian stimulation for in vitro fertilization.

Exclusion Criteria:

* women who underwent ovarian stimulation for cryopreservation in the presence of neoplastic disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with primary or secondary infertility who underwent ovarian stimulation for in vitro fertilization in our centre.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
number of total and mature (MII) oocytes | 10 months
  the number of total and mature (MII) oocytes retrieved during the pick up.

SECONDARY OUTCOMES:
duration of stimulation | 10 months
  the number of days since the administration of rFSH o corifollitropina alfa until the administration of hCG
ovarian sensitivity index or OSI | 10 months
  OSI was calculated dividing the total administered FSH dose by the number of retrieved oocytes
pregnancy rate | 10 months
  the number of positive pregnancy tests with the evidence of an embyo with cardiac activity.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Depalo, MD, Study Director — U.O.S. Procreazione Medicalmente Assistita e Congelamento Gameti, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Bari, Italy

REFERENCES:
- [Result] La Marca A, Papaleo E, Grisendi V, Argento C, Giulini S, Volpe A. Development of a nomogram based on markers of ovarian reserve for the individualisation of the follicle-stimulating hormone starting dose in in vitro fertilisation cycles. BJOG. 2012 Sep;119(10):1171-9. doi: 10.1111/j.1471-0528.2012.03412.x. Epub 2012 Jul 17. PMID 22805536
- [Result] Singh N, Bahadur A, Malhotra N, Kalaivani M, Mittal S. Prospective analysis of ovarian reserve markers as determinant in response to controlled ovarian stimulation in women undergoing IVF cycles in low resource setting in India. Arch Gynecol Obstet. 2013 Sep;288(3):697-703. doi: 10.1007/s00404-013-2802-3. Epub 2013 Mar 26. PMID 23529683
- [Result] Arce JC, La Marca A, Mirner Klein B, Nyboe Andersen A, Fleming R. Antimullerian hormone in gonadotropin releasing-hormone antagonist cycles: prediction of ovarian response and cumulative treatment outcome in good-prognosis patients. Fertil Steril. 2013 May;99(6):1644-53. doi: 10.1016/j.fertnstert.2012.12.048. Epub 2013 Feb 5. PMID 23394782
- [Result] Andersen AN, Witjes H, Gordon K, Mannaerts B; Xpect investigators. Predictive factors of ovarian response and clinical outcome after IVF/ICSI following a rFSH/GnRH antagonist protocol with or without oral contraceptive pre-treatment. Hum Reprod. 2011 Dec;26(12):3413-23. doi: 10.1093/humrep/der318. Epub 2011 Sep 27. PMID 21954280
- [Result] Lan VT, Linh NK, Tuong HM, Wong PC, Howles CM. Anti-Mullerian hormone versus antral follicle count for defining the starting dose of FSH. Reprod Biomed Online. 2013 Oct;27(4):390-9. doi: 10.1016/j.rbmo.2013.07.008. Epub 2013 Jul 23. PMID 23953069